CLINICAL TRIAL: NCT07079202
Title: EFFECT OF KINETIC CONTROL RETRAINING ON ELECTROMYOGRAPHIC ACTIVITY OF TRUNK MUSCLES IN PATIENTS WITH LUMBOSACRAL RADICULOPATHY.
Brief Title: Effect of Kinetic Control in Lumbosacral Radiculopathy.
Acronym: KC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Madonna Maher Ezzat Yassa (Other)
Responsible Party: Sponsor-Investigator, Madonna Maher Ezzat Yassa, Teaching Assistant, Nahda University
Organization: Nahda University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004918
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: LUMBOSACRAL RADICULOPATHY; Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinetic control (Experimental): This group received kinetic control retraining protocol in addition to conventional physical therapy. ( TENS, hot backs, Ultrasound,Nerve mobilization ) three sessions per week for 6 weeks.
  Interventions: Other: kinetic control
- Conventional physical therapy (Active Comparator): This group received only conventional physical therapy. ( TENS, hot backs, Ultrasound, Nerve mobilization ) three sessions per week for 6 weeks.
  Interventions: Other: Conventional physical therapy.

INTERVENTIONS:
Other: kinetic control — Kinetic Control uses the Movement Control Rating System based on motor tests, the purpose of which is to identify the place and direction of uncontrolled movements and exercises to re-educate motor control
  Arms: Kinetic control
Other: Conventional physical therapy. — This group received only conventional physical therapy. ( TENS, hot backs, Ultrasound,Nerve mobilization ) three sessions per week for 6 weeks.
  Arms: Conventional physical therapy

SUMMARY:
-This study would answer the following question: Is there an effect of kinetic control retraining on electromyographic activity of trunk and lumbar proprioception in patients with lumbosacral radiculopathy?

The aims of this study are:

1. To investigate the effect of kinetic control retraining on electromyographic activity of trunk in patients with lumbosacral radiculopathy
2. To investigate the effect of kinetic control retraining on lumbar proprioception in patients with lumbosacral radiculopathy.
3. To investigate the effect of kinetic control retraining on trunk Range of motion (ROM) in patients with lumbosacral radiculopathy.
4. To investigate the effect of kinetic control retraining on pain intensity in patients with lumbosacral radiculopathy. 5 -To investigate the effect of kinetic control retraining on functional disability in patients with lumbosacral radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be from both sexes.
2. The age of patients will range from 35- 50 years old.
3. The Body Mass Index (BMI) of patients will be less than 30Kg/m2
4. All patients represent chronic low back pain (at least 3 months).
5. Patients with unilateral lumbosacral radiculopathy (L4-5, L5-S1) due to Posterolateral disc prolapse.
6. Patients have been diagnosed by MRI.
7. Patients with sufficient cognitive abilities that enables them to understand and follow instructions (Mini-Mental State Examination (MMSE) scale >24).

Exclusion Criteria:

1. Previous spinal surgeries
2. Another Causes of the lumbosacral radiculopathy
3. Pain that persists less than 3 months
4. Spinal tumors
5. Lumbar instability due to structural problems, for example: ligament tear or spondylolythesis.
6. Cognitive impairment (a score less than 24 according to MMSE).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-17 (Estimated); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
ELECTROMYOGRAPHIC ACTIVITY OF TRUNK MUSCLES | 6 Weeks

SECONDARY OUTCOMES:
lumbar proprioception | 6 Weeks
Pain intensity level | 6 weeks
Trunk Rang Of Motion | 6 Weeks
Functional disability level | 6 Weeks